CLINICAL TRIAL: NCT07243275
Title: Comparing the Efficacy of SYSTANE® PRO to MIEBO™ for the Treatment of Dry Eye Disease
Brief Title: SYSTANE® PRO vs. MIEBO™ in Dry Eye Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Anna Tichenor, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28245
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — perfluorohexyl-octan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SYSTANE® PRO (Active Comparator): SYSTANE® PRO is a preservative free artificial tear with a unique triple action formula that contains hyaluronate, nano-sized lipids, and HP-Guar.
  Interventions: Drug: SYSTANE® PRO
- MIEBO™ (Perfluorohexyloctane, PFHO) (Active Comparator): Perfluorohexyloctane (PFHO) ophthalmic solution, which is marketed in the United States as MIEBO™ (Bausch + Lomb; Rochester, NY, USA) is a preservative-free eye drop.
  Interventions: Drug: MIEBO™ (Perfluorohexyloctane, PFHO)

INTERVENTIONS:
Drug: SYSTANE® PRO — SYSTANE® PRO is a preservative free artificial tear with a unique triple action formula that contains hyaluronate, nano-sized lipids, and HP-Guar.
  Arms: SYSTANE® PRO
Drug: MIEBO™ (Perfluorohexyloctane, PFHO) — Perfluorohexyloctane (PFHO) ophthalmic solution, which is marketed in the United States as MIEBO™ (Bausch + Lomb; Rochester, NY, USA) is a preservative-free eye drop.
  Arms: MIEBO™ (Perfluorohexyloctane, PFHO)

SUMMARY:
This is a prospective, randomized, double-masked, multi-site clinical trial designed to compare the efficacy of SYSTANE® PRO (Alcon Laboratories, Inc.) to MIEBO™ (Bausch + Lomb) in treating symptoms of evaporative dry eye disease (DED). The primary goal is to determine whether SYSTANE® PRO is non-inferior to MIEBO™ after one month of treatment, based on change in Ocular Surface Disease Index (OSDI) scores.

ELIGIBILITY:
Inclusion Criteria:

* Adults>=18 years of age
* Corrected visual acuity of 20/100 or better in both eyes
* Ocular Surface Disease Index [OSDI] scores between 23 and 50 units [inclusive]
* Tear break up time score of <=5 seconds in both eyes
* Schirmer I test (without anesthesia) >=5 mm in both eyes

Exclusion Criteria:

* Discontinue contact lens wear starting 7 days prior and throughout the study
* Artificial tears and warm compresses should not be used for at least one week prior to enrollment and throughout the study
* Systemic health conditions that are known to alter tear film physiology(e.g., primary and secondary Sjogren's syndrome)
* History of ocular surgery within the past 12 months
* History of severe ocular trauma, active ocular infection or inflammation, have ever used Accutane or are currently using ocular medications.
* Women who are pregnant or breast feeding(self report)
* Subjects with a condition or in a situation, which in the investigator's opinion, may put the subject at significant rist, may confound the study results, or may significantly interfere with their participation in the study
* Subjects will not be allowed to use any other topical eye drops or other dry eye treatments beyond their assignment during the study
* Participants in clinical trial or study using a device, topical, or oral therapeutic in the past 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
OSDI Scores | Between group difference at 1 month
  Between-group difference in mean change from baseline in Ocular Surface Disease Index (OSDI) Scores at the 1-month visit (0-100 scale).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Eye Research Foundation, Newport Beach, California
  - Indiana Universtiy School of Optometry, Bloomington, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No